CLINICAL TRIAL: NCT03745235
Title: A Randomized Controlled Study Comparing the Influence of a Mindfulness-based Stress Reduction Program vs. Routine Management on Psychological Variables and Biological Markers Related to Immuno-inflammation Associated With Psychological Stress in Caregivers of Patients With Severe Psychiatric Disorders.
Brief Title: A Study Comparing the Influence of a Mindfulness-based Stress Reduction Program vs. Routine Management on Psychological Variables and Biological Markers Related to Immuno-inflammation Associated With Psychological Stress in Caregivers of Patients With Severe Psychiatric Disorders
Acronym: MindInfCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because of the Covid pandemic, group meditation could not be carried out and was not repeated in the study.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Chauvet-Gelinier UNAFAM 2017
Record Dates: First submitted 2018-10-25; First posted 2018-11-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Psychiatry; Caregivers; Mindfulness
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Mindfulness" group (Experimental)
  Interventions: Other: stress reduction program based on mindfulness; Biological: venipunctures; Other: psychometric questionnaires
- Control group (Other): Treatment as Usual
  Interventions: Biological: venipunctures; Other: psychometric questionnaires

INTERVENTIONS:
Other: stress reduction program based on mindfulness — a two and a half hour session per week for 8 weeks
  Arms: "Mindfulness" group
Biological: venipunctures — 1 dry tube of 5 ml and 5 heparinized tubes of 6 ml taken at inclusion, at 3 months and at 12 months
Other: psychometric questionnaires — * Cohen PSS' perceived stress scale
  * Beck's anxiety and depression questionnaires
  * Watson's affectivity questionnaire, positive affect and negative affect schedule
  * optimism questionnaire, Life Orientation Test LOT-R by Sheier and Carver
  * IN-OUT DASQ dispositional affective style questionnaire

SUMMARY:
The objective of this project is to study the influence of mindfulness meditation on psychological health (stress level, affects, emotions) and physical health parameters (rate of inflammatory markers in the blood, activity of white blood cells involved in immuno-inflammation) in caregivers of people with psychiatric disorders. This study will provide the objective scientific data required for the development of mindfulness meditation programs for psychiatric caregivers.

80 participants will be randomly assigned to one of the following two groups:

* 40 participants in the "Mindfulness" group who will attend mindfulness meditation sessions in addition to their standard follow-up
* 40 participants in the "Control" group who will have a standard follow-up The duration of participation is 12 months and includes 3 visits and 8 mindfulness-based meditation sessions for the "Mindfulness" group.

ELIGIBILITY:
Inclusion Criteria:

* patient who has given oral consent
* adult patient
* a caregiver of a person with a severe psychiatric disorder (schizophrenia, recurrent depression, bipolar disorder, obsessive-compulsive disorder)

Exclusion Criteria:

* protected adult
* patient not affiliated to the national health insurance system
* pregnant, parturient or breastfeeding woman
* person suffering from a severe psychiatric disorder indicating a state of decompensated stress (with risk of associated biological inflammatory disturbances)
* person suffering from an inflammatory disease (autoimmune, infectious, neoplastic, cardio-vascular pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
measurement of inflammation by analysis of US-CRP blood levels | Change from Baseline US-CRP blood levels at 3 and 12 months
measurement of inflammation by analysis of IL-6 blood levels | Change from Baseline IL-6 blood levels at 3 and 12 months
measurement of lymphocyte activity Th1 Th2 Th17 Treg | Change from Baseline lymphocytes activity Th1 Th2 Th17 Treg at 3 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No